CLINICAL TRIAL: NCT07372937
Title: Investigating Neural Correlates of Gait Abnormalities in Patients With Cerebral Small Vessel Disease
Brief Title: Neural Correlates (EEG and fMRI) of Gait in Small Vessel Disease
Acronym: doesn't exist
Status: Not yet recruiting | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Hadeer Samir Ahmed Hamada, Assistant lecturer of neurology, MD candidate , Ain Shams University, Ain Shams University
Other Study IDs: FMASU132/2025
Record Dates: First submitted 2026-01-20; First posted 2026-01-28 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Cerebral Small Vessel Disease
Keywords: Gait Disturbances, Vascular cognitive impairment; gait disturbances; vascular cognitive impairment
MeSH Terms: conditions — Cerebral Small Vessel Diseases; Mobility Limitation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Controls: Age matched adults with no neurological disorders or gait impairments and normal MRI findings. Participants will undergo the same clinical, EEG, and MRI assessments as the patient group.
  Interventions: Other: No Intervention: Observational
- SVD Patients: dults aged 50 years or older diagnosed with cerebral small vessel disease (SVD) showing gait disturbance confirmed by MRI (Fazekas score 2-3). Participants will undergo clinical assessment, EEG, and functional MRI.
  Interventions: Other: No Intervention: Observational

INTERVENTIONS:
Other: No Intervention: Observational — no intervention

SUMMARY:
What is the purpose of this study? This observational study is being done to understand how cerebral small vessel disease (SVD) affects walking and balance. SVD is a common brain condition in older adults that damages small blood vessels. It can lead to problems with movement, thinking, and memory. The researchers want to find out how changes in brain activity and connectivity contribute to walking difficulties in people with SVD.

Why is this study important? Walking and balance problems increase the risk of falls and loss of independence. By studying brain activity during walking-related tasks, researchers hope to identify patterns that explain why these problems happen. This knowledge could help develop better rehabilitation methods in the future.

Who can participate? Adults over 50 years old with cerebral small vessel disease and gradual gait problems may be eligible. Healthy adults of similar age without neurological problems may also take part as control participants.

What will happen in this study?

Participants will:

Complete walking, balance, and cognitive tests such as the Timed Up and Go, Berg Balance Scale, and Montreal Cognitive Assessment.

Undergo brain imaging (MRI) to confirm the diagnosis and study brain structure and function.

Have an EEG recording while resting and while watching short videos showing walking and turning movements.

A smaller group will also undergo functional MRI (fMRI) while watching the same videos.

The MRI and EEG results will be analyzed to see how brain networks involved in movement and balance differ between patients and healthy adults.

How long will the study take? The study will take about two years to complete. Each participant's visit will last approximately two to three hours in total.

What are the possible benefits? There may be no direct benefit to participants. However, this study may help researchers understand how small vessel disease affects brain function related to walking, which may improve care for future patients.

DETAILED DESCRIPTION:
Cerebral small vessel disease (SVD) is a common cause of walking and balance problems in older adults. These problems are often not explained by muscle weakness alone. They are believed to result from changes in how different parts of the brain communicate and coordinate movement.

This study will explore how brain network function is affected in people with SVD who experience gait difficulties. To do this, two safe and non-invasive techniques will be used:

Functional MRI (fMRI): to identify which brain areas become active when participants watch videos that simulate walking and turning.

Electroencephalography (EEG): to measure brain waves and the timing of brain activity while watching the same gait-related videos.

Participants will include 20 patients diagnosed with cerebral small vessel disease and gait problems, and 20 healthy adults of similar age without such problems.

All participants will undergo:

1. Clinical evaluation including walking, balance, and cognitive tests (Timed Up and Go, Berg Balance Scale, and Montreal Cognitive Assessment).
2. Brain MRI to confirm the diagnosis and exclude other causes.
3. Resting and task-based EEG recordings to assess brain connectivity.
4. Functional MRI for a subset of participants to study brain activity patterns related to gait imagery.

Researchers will compare the brain activation and connectivity between patients and healthy participants. They will also look for relationships between imaging findings and clinical test results.

By combining fMRI and EEG findings, this research aims to identify brain networks that are disrupted in people with SVD-related gait problems. Understanding these patterns may lead to better tools for early detection and more targeted rehabilitation approaches to improve walking and prevent falls.

All study procedures will be conducted at the Neurology Department, Ain Shams University Hospitals, Cairo, Egypt.

ELIGIBILITY:
Inclusion Criteria:

* Age 50 years or older.
* Clinical and radiological diagnosis of cerebral small vessel disease (SVD), confirmed by MRI findings such as white matter hyperintensities, lacunes, or microbleeds.
* Fazekas score 2 or 3 on MRI.
* Presence of slowly progressive gait disturbance (e.g., slowness, imbalance, freezing) rather than acute stroke presentation.

  * Ability to give informed consent and cooperate with testing procedures.

Exclusion Criteria:

* Presence of other neurodegenerative disorders (e.g., Parkinson's disease, Alzheimer's disease).
* History of large vessel stroke or intracerebral hemorrhage.
* Contraindications to MRI (e.g., pacemaker, metallic implants, severe claustrophobia).
* Severe cognitive impairment that prevents participation (MoCA <10).
* Musculoskeletal or orthopedic causes of gait disturbance not related to neurological dysfunction.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults aged 50 years or older attending the Neurology outpatient clinics at Ain Shams University Hospitals, including patients with small vessel disease and gait impairment, and healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Functional brain connectivity differences between SVD patients and healthy controls | At baseline (single assessment visit)
  Differences in resting-state and task-based EEG connectivity and fMRI network activation between patients with cerebral small vessel disease and healthy controls. Connectivity will be analyzed using coherence, phase-locking value (PLV), and correlation matrices derived from resting-state fMRI and EEG. The goal is to identify altered cortico-subcortical communication associated with gait impairment.

SECONDARY OUTCOMES:
Correlation between imaging findings and clinical gait performance | At baseline (single assessment visit)
  Evaluate the relationship between EEG/fMRI connectivity parameters and scores on the Timed Up and Go (TUG) test and Berg Balance Scale (BBS) to assess how altered connectivity relates to walking and balance difficulties in SVD.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Hospitals, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
The research team will decide after study completion whether de-identified participant data may be shared.
  Time Frame To be determined after publication. Access Criteria Requests may be directed to the principal investigator and will require approval by the Faculty of Medicine, Ain Shams University.

REFERENCES:
- [Result] Torres-Simon L, Doval S, Nebreda A, Llinas SJ, Marsh EB, Maestu F. Understanding brain function in vascular cognitive impairment and dementia with EEG and MEG: A systematic review. Neuroimage Clin. 2022;35:103040. doi: 10.1016/j.nicl.2022.103040. Epub 2022 May 10. PMID 35653914
- [Result] Su C, Yang X, Wei S, Zhao R. Association of cerebral small vessel disease with gait and balance disorders. Front Aging Neurosci. 2022;14:834496. PMID: 35528672
- [Result] Mele G, Cavaliere C, Alfano V, Orsini M, Salvatore M, Aiello M. Simultaneous EEG-fMRI for Functional Neurological Assessment. Front Neurol. 2019 Aug 13;10:848. doi: 10.3389/fneur.2019.00848. eCollection 2019. PMID 31456735
- [Result] Schulz M, Malherbe C, Cheng B, Thomalla G, Schlemm E. Functional connectivity changes in cerebral small vessel disease - a systematic review of the resting-state MRI literature. BMC Medicine. 2021;19(1):234. PMID: 34521428
- [Result] Sharma B, Wang M, McCreary CR, Camicioli R, Smith EE. Gait and falls in cerebral small vessel disease: a systematic review and meta-analysis. Age Ageing. 2023 Mar 1;52(3):afad011. doi: 10.1093/ageing/afad011. PMID 37000039